CLINICAL TRIAL: NCT03258112
Title: Safety and Efficacy of Catheter Ablation of Idiopathic Ventricular Arrhythmias Arising From Cardiac Outflow Tracts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: I have changed my center and gone to another center
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abo Elhassan Abdel_Rady, M. abo Elhassan, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: electrophysiology
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Ventricular Arrythmia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- catheter ablation (Other): all patients indicated for catheter ablation of RVOT or LVOT ventricular arrhythmia are included in one arm for electrophysiological diagnosis of the origin of arrhythmia then for radiofrequency catheter ablation
  Interventions: Procedure: Radiofrequency cardiac catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency cardiac catheter ablation — procedure used for ablation of ventricular arrhythmia using catheters introduced to target sites percutaneously through venous or arterial systems using radiofrequency power

SUMMARY:
Ventricular arrhythmias arising from cardiac outflow tract affect quality of life and can cause decrease in left ventricular ejection fraction.

Drugs used for treating those arrhytmias may be ineffective or may have side effects.

Radiofrequency catheter ablation can be used safely for treatment of outflow tract arrhythmias.

There are different sites where those ventricular arrhythmias may originates, each site has different electrocardiographic characteristics, different procedural success rates and challenges in localization and ablation.

DETAILED DESCRIPTION:
The right and left ventricular outflow tracts (RVOT/LVOT) are the most common sites of origin for idiopathic ventricular tachycardia (VT) and premature ventricular contractions (PVCs) in patients without structural heart disease.1

Frequent PVCs was associated with PVC-induced cardiomyopathy, and radiofrequency (RF) catheter ablation of frequent PVCs was associated with improvement of left ventricular ejection fraction (LVEF).2

The most common underlying pathophysiological mechanism was identified to be triggered activity and RF catheter ablation treatment is highly effective with low complication rates.1,3 Drug therapy has limited effectiveness (in case β-blockers and calcium-channel blockers) or drug-related side effects ( in case of flecainide, propafenone and amiodarone).4

RF catheter ablation is recommended in cases of high PVC burden associated with decreased LV ejection fraction (LVEF) or in highly symptomatic patients despite optimal drug therapy.3

Although the RVOT is the most common site (about 70-80% of cases) for idiopathic VAs1,5, only few studies have reported on the prevalence and RF catheter ablation of ventricular arrhythmias (VAs) arising from the pulmonary artery (21-46% among the RVOT VAs)6 and even less prevalence is reported in VAs arising from the pulmonary sinus cusps (11%).7

Compared with VAs originating from the RVOT, ablation of LVOT-VAs is more complex and reported to be 12-45% of all idiopathic VAs.8-11 The success rate of ablation of LVOT-VA sites was previously reported to be lower (55-60%) without using antegrade/transseptal approaches.12,4 Rarely, it requires epicardial ablation via the GCV/AIV or subxiphoid puncture.13,14

There are some cases in which RF catheter ablation cannot successfully be performed from either LVOT or RVOT. In such cases the VAs may originate from the LV-summit which is the most common site of idiopathic epicardial VAs from the LVOT region.13

Although most idiopathic VAs originating from the cardiac OTs are suitable targets for endocardial RF catheter ablation, a small percentage of failures in these patients may be because of an inaccessible site of origin from epicardial or intramural septal locations.15The identification, mapping and RF catheter ablation of these idiopathic VAs may be challenging for the electrophysiologist and need special consideration.16

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic RVOT/LVOT ventricular arrhythmias in cases of Frequent (PVCs =10.000/24hours), NSVT, or VT Symptomatic, Associated with LV dysfunction (no explained with any cause other than VAs) or Resistance, patient intolerance or patient refusal of drug therapy

Exclusion Criteria:

* Presence of coronary artery disease, valvular heart disease or any other underlying causes
* arrhythmia not originating from cardiac outflow tracts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
procedural success | 24 hours after the procedure
  success of the procedure in ablation of ventricular arrhythmia with termination of ventricular arrhythmia, absence of induction of arrhythmia and 24 hours electrocardiographic monitoring after the procedure documenting absence of ventricular arrhythmia

SECONDARY OUTCOMES:
Recurrence of ventricular arrhythmia after three months | Three months
  Appearance of symptoms of palpitation and documentation of recurrence of same type of arrhythmia with prolonged electrocardiographic monitoring in case of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abo Elhassan Abdel-Rady, Principal Investigator — Assiut University

REFERENCES:
- [Background] Latchamsetty R, Yokokawa M, Morady F, Kim HM, Mathew S, Tilz R, et al. Multicenter outcomes for catheter ablation of idiopathic premature ventricular complexes. J Am Coll Cardiol EP 2015; 1: 116 - 123
- [Background] Kumagai K. Idiopathic ventricular arrhythmias arising from the left ventricular outflow tract: Tips and tricks. J Arrythmia 2014; 30: 211 - 221
- [Result] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; ESC Scientific Document Group. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J. 2015 Nov 1;36(41):2793-2867. doi: 10.1093/eurheartj/ehv316. Epub 2015 Aug 29. No abstract available. PMID 26320108
- [Result] Wojdyla-Hordynska A, Kowalski O, Hordynski GJ, Dinov B, Sommer P, Hindricks G, Feusette P, Arya A. The effect of radiofrequency catheter ablation of frequent premature ventricular complexes and arrhythmia burden on left ventricular function. Kardiol Pol. 2017;75(7):698-704. doi: 10.5603/KP.a2017.0058. PMID 28708198
- [Result] Pedersen CT, Kay GN, Kalman J, Borggrefe M, Della-Bella P, Dickfeld T, Dorian P, Huikuri H, Kim YH, Knight B, Marchlinski F, Ross D, Sacher F, Sapp J, Shivkumar K, Soejima K, Tada H, Alexander ME, Triedman JK, Yamada T, Kirchhof P, Lip GY, Kuck KH, Mont L, Haines D, Indik J, Dimarco J, Exner D, Iesaka Y, Savelieva I; EP-Europace,UK. EHRA/HRS/APHRS expert consensus on ventricular arrhythmias. Heart Rhythm. 2014 Oct;11(10):e166-96. doi: 10.1016/j.hrthm.2014.07.024. Epub 2014 Aug 30. No abstract available. PMID 25179489
- [Result] Pytkowski M, Maciag A, Sterlinski M, Jankowska A, Kowalik I, Farkowski MM, Kuteszko R, Zajac D, Firek B, Chmielak Z, Szwed H. Novel algorithm for arrhythmogenic focus localization in patients with right ventricular outflow tract arrhythmias. Cardiol J. 2014;21(3):284-92. doi: 10.5603/CJ.a2013.0111. Epub 2013 Aug 30. PMID 23990183
- [Result] Timmermans C, Rodriguez LM, Crijns HJ, Moorman AF, Wellens HJ. Idiopathic left bundle-branch block-shaped ventricular tachycardia may originate above the pulmonary valve. Circulation. 2003 Oct 21;108(16):1960-7. doi: 10.1161/01.CIR.0000095026.19339.BB. Epub 2003 Oct 6. PMID 14530199
- [Result] Liao Z, Zhan X, Wu S, Xue Y, Fang X, Liao H, Deng H, Liang Y, Wei W, Liu Y, Ouyang F. Idiopathic Ventricular Arrhythmias Originating From the Pulmonary Sinus Cusp: Prevalence, Electrocardiographic/Electrophysiological Characteristics, and Catheter Ablation. J Am Coll Cardiol. 2015 Dec 15;66(23):2633-2644. doi: 10.1016/j.jacc.2015.09.094. PMID 26670064
- [Result] Kamioka M, Mathew S, Lin T, Metzner A, Rillig A, Deiss S, Rausch P, Lemes C, Makimoto H, Hu H, Liang D, Wissner E, Tilz RR, Kuck KH, Ouyang F. Electrophysiological and electrocardiographic predictors of ventricular arrhythmias originating from the left ventricular outflow tract within and below the coronary sinus cusps. Clin Res Cardiol. 2015 Jul;104(7):544-54. doi: 10.1007/s00392-015-0817-4. Epub 2015 Jan 30. PMID 25633492
- [Result] Yamada T, Litovsky SH, Kay GN. The left ventricular ostium: an anatomic concept relevant to idiopathic ventricular arrhythmias. Circ Arrhythm Electrophysiol. 2008 Dec;1(5):396-404. doi: 10.1161/CIRCEP.108.795948. No abstract available. PMID 19808434
- [Result] Ouyang F, Mathew S, Wu S, Kamioka M, Metzner A, Xue Y, Ju W, Yang B, Zhan X, Rillig A, Lin T, Rausch P, Deiss S, Lemes C, Tonnis T, Wissner E, Tilz RR, Kuck KH, Chen M. Ventricular arrhythmias arising from the left ventricular outflow tract below the aortic sinus cusps: mapping and catheter ablation via transseptal approach and electrocardiographic characteristics. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):445-55. doi: 10.1161/CIRCEP.114.001690. Epub 2014 May 2. PMID 24795340
- [Result] Ouyang F, Fotuhi P, Ho SY, Hebe J, Volkmer M, Goya M, Burns M, Antz M, Ernst S, Cappato R, Kuck KH. Repetitive monomorphic ventricular tachycardia originating from the aortic sinus cusp: electrocardiographic characterization for guiding catheter ablation. J Am Coll Cardiol. 2002 Feb 6;39(3):500-8. doi: 10.1016/s0735-1097(01)01767-3. PMID 11823089
- [Result] Yamada T, McElderry HT, Doppalapudi H, Okada T, Murakami Y, Yoshida Y, Yoshida N, Inden Y, Murohara T, Plumb VJ, Kay GN. Idiopathic ventricular arrhythmias originating from the left ventricular summit: anatomic concepts relevant to ablation. Circ Arrhythm Electrophysiol. 2010 Dec;3(6):616-23. doi: 10.1161/CIRCEP.110.939744. Epub 2010 Sep 20. PMID 20855374
- [Result] Ouyang F, Bansch D, Schaumann A, Ernst S, Linder C, Falk P, Hachiya H, Kuck KH, Antz M. Catheter ablation of subepicardial ventricular tachycardia using electroanatomic mapping. Herz. 2003 Nov;28(7):591-7. doi: 10.1007/s00059-003-2494-8. PMID 14689119
- [Result] Yokokawa M, Good E, Chugh A, Pelosi F Jr, Crawford T, Jongnarangsin K, Latchamsetty R, Oral H, Morady F, Bogun F. Intramural idiopathic ventricular arrhythmias originating in the intraventricular septum: mapping and ablation. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):258-63. doi: 10.1161/CIRCEP.111.967257. Epub 2012 Mar 9. PMID 22407415
- [Result] Heeger CH, Hayashi K, Kuck KH, Ouyang F. Catheter Ablation of Idiopathic Ventricular Arrhythmias Arising From the Cardiac Outflow Tracts - Recent Insights and Techniques for the Successful Treatment of Common and Challenging Cases. Circ J. 2016 Apr 25;80(5):1073-86. doi: 10.1253/circj.CJ-16-0293. Epub 2016 Apr 13. PMID 27074752